CLINICAL TRIAL: NCT03993093
Title: AIDS Defining Opportunistic Infections in Naive HIV Cases
Brief Title: Prevalence of HIV +ve Cases With AIDS Defining Opportunistic Infections Among ART Naive Patients Attending ART Centre
Acronym: ADC
Status: Completed | Type: Observational
Sponsor: Singh, Ranjan Kumar, M.D. (Individual)
Responsible Party: Principal Investigator, Ranjan Kumar Singh, Physician, cum nodal officer, ART centre Khagaria, Singh, Ranjan Kumar, M.D.
Other Study IDs: SinghRK1
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: HIV Infections; Tuberculosis; Candidiasis, Esophageal; Cryptococcosis; Leishmaniasis; Toxoplasmosis
Keywords: HIV; Opportunistic infection; CD4+ T cells; AIDS defining condition
MeSH Terms: conditions — HIV Infections; Tuberculosis; Candidiasis; Cryptococcosis; Leishmaniasis; Toxoplasmosis; Opportunistic Infections | interventions — CD4 Lymphocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV with OIs: Treatment naive HIV patients with OIs
  Interventions: Other: CD4 cell count

INTERVENTIONS:
Other: CD4 cell count — CD4 cell count from treatment naive HIV patients

SUMMARY:
HIV patients are likely to suffer from opportunistic infections, in absence of highly active retroviral therapy. This happens due to lack of awareness of HIV status among patients or unresponsive to anti retroviral drugs. This study is for the prevalence of AIDS defining OIs among treatment naive HIV patients.

DETAILED DESCRIPTION:
Oppotunistic infections (OIs) happen in persons with weakened immune system. HIV patients, who remain untreated due to lack of knowledge of existing HIV infections, often get OIs. HIV patients with AIDS defining OIs fall into stage 3 of HIV illness. Prevalence of OIs in resource poor settings are tuberculosis (pulmonary and extra pulmonary), toxoplasmosis, cryptococcosis, and oesophageal candidiasis. There are a few data to show AIDS defining OIs in treatment naïve HIV patients. Incidence of OIs among HIV patients in United States, and Canada between 2000 to 2019 was 9%. Leading OIs were peumocystis Jiroveci, oesophageal candidiasis and disseminated MAC or M. kansassi.

Minimal diagnoses at poor settings can be made by observation of symptoms, use of microscope, imaging and diagnostic therapy.

ELIGIBILITY:
Inclusion Criteria:

• HAART naïve HIV patient

Exclusion Criteria:

* Patients died during screening
* Transferred in HIV patients

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Antiretroviral treatment naive HIV patients
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of AIDS defining OIs | Six months
  Calculate number of total HIV patients with or without opportunistic infections (n). Again calculate no of HIV patients with opportunistic infections (n1). Then calculate prevalence of HIV +ve patients with opportunistic infections by applying formula n1/n x100.

SECONDARY OUTCOMES:
Compare CD4 cell in cases of HIV with OIs with CD4 cell of HIV patients without OIs | Six months
  Find out CD4 cell counts (cells /μL) of HIV patients with CD4 cell counts (cells/μL) of HIV patients without OIs. By calculating mean/SD of CD4 cells in both groups, comparison by chi square test would be done.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan K Singh, M.D., Principal Investigator — Singh, Ranjan Kumar
Locations (1):
- ART centre, Sadar Hospital, Khagaria, Bihar, India